CLINICAL TRIAL: NCT04278508
Title: Is There an Association Between Low Serum Progesterone on the Day of Frozen-thawed Embryo Transfer and a Reduced Clinical Pregnancy Rate After an Artificial Endometrial Preparation: A Randomized Control Trial
Brief Title: Serum Progesterone on the Day of Thawed Embryo Transfer and Pregnancy Rate After an Artificial Endometrial Preparation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 0155-19-HYMC
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: IVF
MeSH Terms: interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): P < 10.0 ng/ml with increasing P dosage from 800 mg to 1200 mg daily from the FET day.
  Interventions: Drug: Progesterone
- Group B (Active Comparator): P < 10.0 ng/ml without change in drug regimen.
  Interventions: Drug: Progesterone
- Group C (Active Comparator): P ≥ 10.0 ng/ml without change in drug regimen.
  Interventions: Drug: Progesterone

INTERVENTIONS:
Drug: Progesterone — To determine if different serum P levels on FET day are associated with different clinical pregnancy rates (CPR)

SUMMARY:
To determine if different serum Progesterone levels on FET day are associated with different clinical pregnancy rates (CPR), and if increasing dosage of vaginal Progesterone in cases of lower serum Progesterone level on FET day can be either beneficial or detrimental regarding the CPR.

DETAILED DESCRIPTION:
Over the past decade, the use of frozen-thawed embryo transfer (FET) has risen around the globe. There is no consensus which mode of FET is superior, either natural cycle (NC) or artificial cycle (AC) with hormonal replacement therapy (HRT). The latter has become more and more popular because it allows more flexibility in timing of FET and it requires fewer visits for monitoring before the transfer. AC also has the advantage of a more precise control of progesterone (P) exposure, which is of utmost importance for controlling the window of implantation between the embryo and the endometrium. Although FET in AC give excellent results, there is still a need for improvement, as the ideal dose is not individualized to a patient's characteristics and serum P required for optimal cycle outcome haven't been established.

Retrospective studies about P levels on the day of FET in AC cycles showed contradictory results regarding cycle outcomes. Several studies showed that a lower P levels on FET day, or one day prior, are associated with lower clinical pregnancy rate (CPR) or live birth rate (LBR), whereas one study showed that women with higher P on FET day were having lower LBRs. Recently, a prospective study showed that serum P level < 9.2 ng/ml on the day of FET in oocyte reception cycles was associated with a significant lower ongoing pregnancy rate. Considering these previous studies, we wanted to determine if different serum P levels on FET day are associated with different CPR, and if increasing dosage of vaginal P in cases of lower serum P level on FET day can be either beneficial or detrimental.

ELIGIBILITY:
Inclusion Criteria:

* women between age 18-38 undergoing FET in AC
* with body mass index (BMI) < 35 kg/m2
* a triple layer endometrium >6.5 mm after exogenous estrogen administration
* 1-2 good quality day 3 or 5 FET.

Exclusion Criteria:

* women with recurrent pregnancy losses (e.g. 2 abortions beyond 12th week or 3 abortions before 12th week)
* recurrent implantation failure (e.g. unsuccessful implantation of ≥4 good quality embryos)
* severe male factor (sperm concentration <5 million/ml), or presence of hydrosalpinx.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 38 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 1 Year per patient
  Clinical pregnancy rate according to the presence of pregnancy sac on week 6-7 US.

SECONDARY OUTCOMES:
Laboratory end other long term outcomes | 1 Year per patient
  chemical pregnancy rate, miscarriage rate, and live birth rates.

CONTACTS AND LOCATIONS:
Overall Officials: Einat Shalom-Paz, Prof., Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel